CLINICAL TRIAL: NCT04123210
Title: Development of 13C-Retinol Isotope Dilution Techniques
Brief Title: Estimating Average Vitamin A Requirements in Indonesian and American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-2007-0324; A074600 (Other: UW, Madison); AG&LSC/NUTRITIONAL SCI/NUTRITI (Other: UW, Madison)
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Vitamin A Deficiency
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Intervention Model Description: Parallel assignment to 0 or 525 micrograms supplemental vitamin A/day (Indonesia) or 0, 175 or 525 micrograms supplemental vitamin A/day (USA).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants blinded (Indonesian), double blinded (USA)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin A supplement (Experimental): Subjects receive a vitamin A supplement containing 175 or 525 micrograms of vitamin A as retinyl palmitate daily
  Interventions: Dietary Supplement: Vitamin A supplement
- Placebo (Placebo Comparator): Subjects receive an oil placebo containing no vitamin A
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin A supplement
  Arms: Vitamin A supplement
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Women of reproductive age had their vitamin A stores estimated by retinol isotope dilution and then were given vitamin A supplements near the US vitamin A RDA or placebo for 42(USA) or 60 (Indonesia) days, after which retinol isotope dilution was repeated and the change in vitamin A stores was determined in each group to estimate how much vitamin A is needed to maintain nutrient balance in these women.

ELIGIBILITY:
Inclusion Criteria:

* Normal nutritional status (BMI 18.5-25)

Exclusion Criteria:

* Significant clinical illness

Ages: 19 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2008-03-17 (Actual); Primary Completion 2009-05-05 (Actual); Study Completion 2009-05-05 (Actual)

PRIMARY OUTCOMES:
Total body vitamin A stores (micromoles of vitamin A) | Baseline and after 42 to 60 days
  Change in total body stores of vitamin A before and after intervention, measured by retinol isotope dilution
Total vitamin A liver reserves (micromoles vitamin A per gram liver) | Baseline and after 42 to 60 days
  Change in total liver reserves of vitamin A before and after intervention, measured by retinol isotope dilution

CONTACTS AND LOCATIONS:
Overall Officials: Sherry A Tanumihardjo, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- University of Wisconsin - Madison, Madison, Wisconsin, United States
- Pusat Teknologi Terapan Kesehatan dan Epidemiologi Klinik, Bogor, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheftel J, Valentine AR, Hull AK, Fadjarwati T, Gannon BM, Davis CR, Tanumihardjo SA. Findings in 3 clinical trials challenge the accuracy of the Institute of Medicine's estimated average requirements for vitamin A in children and women. Am J Clin Nutr. 2021 May 8;113(5):1322-1331. doi: 10.1093/ajcn/nqaa132. PMID 32492125